CLINICAL TRIAL: NCT07060508
Title: Safety and Efficacy of L9LS, a Human Monoclonal Antibody Against Plasmodium Falciparum, in a Randomized, Double-Blind, Placebo-Controlled Trial of Women of Childbearing Potential (WOCBP) in Mali
Brief Title: L9LS in Women of Childbearing Potential in Mali
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Malaria Research and Training Center, Bamako, Mali (Other); University of the Sciences, Techniques and Technologies of Bamako (Other); Faculté de Médecine Pharmacie d'Odontostomatologie (FMOS) (Unknown); University of Washington (Other); Harvard School of Public Health (HSPH) (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: L9LS in WOCBP
Record Dates: First submitted 2025-06-10; First posted 2025-07-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- L9LS in healthy Malian WOCBP (Experimental)
  Interventions: Biological: Single dose of 1800 mg L9LS SC
- Placebo in healthy Malian WOCBP (Placebo Comparator)
  Interventions: Other: Placebo
- L9LS in healthy Malian adult males (Experimental)
  Interventions: Biological: Single dose of 1800 mg L9LS SC

INTERVENTIONS:
Biological: Single dose of 1800 mg L9LS SC — A human monoclonal antibody to protect against Plasmodium falciparum.
  Arms: L9LS in healthy Malian WOCBP; L9LS in healthy Malian adult males
Other: Placebo — Normal saline
  Arms: Placebo in healthy Malian WOCBP

SUMMARY:
Safety and Efficacy of L9LS, a Human Monoclonal Antibody Against Plasmodium falciparum, in a Randomized, Double-Blind, Placebo-Controlled Trial of Women of Childbearing Potential (WOCBP) in Mali

DETAILED DESCRIPTION:
This is a phase 2 trial evaluating the safety and tolerability of a 1-time subcutaneous (SC) administration of L9LS, as well as its protective efficacy against naturally occurring Plasmodium falciparum (Pf) infection over a 6-month malaria season. The primary study hypothesis is that L9LS will be safe and protective against malaria infection. As a secondary objective, the efficacy of L9LS among female participants of childbearing potential within three body weight strata will be compared to placebo. Before study agent administration, all participants will be given artemether-lumefantrine (AL) to clear any preexisting Pf blood stage infection.

This is a randomized, double-blind, placebo-controlled study mainly in WOCBP, weight-stratified (N=270 total), with 2 treatment arms: L9LS 1800 mg SC (n=180) and placebo (n=90) to assess safety and protective efficacy of L9LS. A separate open label male only arm (n=20) will assess sex-differences in the pharmacokinetics (PK) of L9LS at a dose of 1800 mg SC. Male participants will be enrolled during the same time period as the WOCBP arm.

Participants will receive the study agent and be followed at visits on study Days 1, 3, 7, 14, 21, and 28 days later, and once every 2 weeks thereafter through 24 weeks. Primary study assessments include physical examination, blood collection for identification of Pf infection and other research laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged ≥18 and ≤49 years and weighing ≥ 45.0 and ≤ 90.0 kg.
2. Males aged ≥18 and ≤49 years (no weight restrictions).
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. In good general health and without clinically significant medical history.
5. Able to provide informed consent.
6. Willing to have blood samples and data stored for future research.
7. Resides in or near Kalifabougou, Faladje, or Torodo, Mali, and available for the duration of the study.
8. Females of childbearing potential must be willing to use reliable contraception from 21 days prior to study Day 0 through the final study visit as described below.

   1. Reliable methods of birth control include 1 of the following: confirmed pharmacologic contraceptives via parenteral delivery or intrauterine or implantable device.

Exclusion Criteria:

1. Pregnancy, as determined by a positive urine or serum beta-human choriogonadotropin (β hCG) test (if female).
2. Currently breastfeeding.
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol.
4. Study comprehension examination score of <80% correct or per investigator discretion.
5. Hemoglobin, WBC, absolute neutrophil, or platelet count outside the local laboratory-defined limits of normal. (Participants may be included at the investigator's discretion for "not clinically significant" values.)
6. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal. (Participants may be included at the investigator's discretion for "not clinically significant" values.)
7. Infected with HIV, hepatitis C virus (HCV), or hepatitis B virus (HBV).
8. Known or documented sickle cell disease by history. (Note: Known sickle cell trait is NOT exclusionary.)
9. Clinically significant abnormal electrocardiogram (ECG; QTc >460 or other significant abnormal findings, including unexplained tachycardia or bradycardia).
10. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
11. Receipt of any investigational product within the past 30 days.
12. Participation or planned participation in an interventional trial with an investigational product until the last required protocol visit. [Note: Past, current, or planned participation in observational studies is NOT exclusionary; participation in the placebo arm of the Mali adult CIS43LS MAb trial (ClinicalTrials.gov Identifier: NCT04329104) or the placebo arm of the Mali adult L9LS Mab trial (ClinicalTrials.gov Identifier: NCT05816330) is NOT exclusionary.]
13. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
14. History of a severe allergic reaction or anaphylaxis.
15. Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years).
16. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, or autoimmune thrombocytopenia.
17. Salivary gland disorder diagnosed by a doctor (e.g., parotitis, sialadenitis, sialolithiasis, salivary gland tumors).
18. Known immunodeficiency syndrome.
19. Known asplenia or functional asplenia.
20. Use of chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of day 0.
21. Receipt of a live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks prior to study agent administration.
22. Receipt of immunoglobulins and/or blood products within the past 6 months.
23. Previous receipt of an investigational malaria vaccine or MAb in the last 5 years.
24. Known allergies or contraindication against artemether lumefantrine.
25. Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or render the participant unable to comply with the protocol.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of local and systemic adverse events (AEs) | Days 0, 1, 3, and 7.
  Occurring within 7 days after the administration of study agent
Severity of local and systemic adverse events (AEs) | Days 0, 1, 3, and 7.
  Occurring within 7 days after the administration of study agent
Incidence of laboratory abnormalities | Days 7 and 14.
  Occurring within 14 days after the administration of study agent
Number of participants with treatment-related laboratory adverse events | Days 7 and 14.
  Occurring within 14 days after the administration of study agent
Pf blood-stage infection as detected by microscopic examination of thick blood smear | Once every 2 weeks post injection through 24 weeks.

SECONDARY OUTCOMES:
Pf blood-stage infection as detected by thick blood smear and RT-PCR | Blood smear once every 2 weeks post injection through 24 weeks.
  For 24 weeks after administration of study agent.
Concentration of L9LS in sera of recipients. | Through 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Crompton, MD, MPH, Principal Investigator — National Institutes of Health (NIH); Kassoum Kayentao, MD, MPH, PhD, Principal Investigator — Faculté de Médecine Pharmacie d'Odontostomatologie (FMOS)
Locations (3):
- Mali (3):
  - Faladje MRTC Clinic, Faladié, Koulikoro
  - Kalifabougou MRTC Clinic, Kalifabougou, Koulikoro
  - Torodo MRTC Clinic, Torodo, Koulikoro

IPD SHARING:
Plan to Share IPD: Yes
Human data generated in this study for future research will be shared as follows:
  * De-identified or identified data with approved outside collaborators under appropriate agreements.
  * De-identified results or data in publication and/or public presentations.
Supporting Information: Study Protocol
Time Frame: Data will be shared at the time of publication or shortly thereafter.
Access Criteria: Data from this study may be requested from other researchers indefinitely after the completion of the primary endpoint by contacting the Laboratory of Immunogenetics at NIH